CLINICAL TRIAL: NCT02510885
Title: Spectral Domain-Optical Coherence Tomography Angiography of Retinal Diseases
Brief Title: SD-OCT Angiography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to COVID-19
Sponsor: Duke University (Other)
Collaborators: Optovue (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00063777
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Neovascular Age-related Macular Degeneration; Age-related Macular Degeneration; Diabetic Retinopathy; Retinal Vein Occlusion; Diabetic Macular Edema
Keywords: neovascular age-related macular degeneration; age-related macular degeneration; diabetic retinopathy; SD-OCT; Angiography; diabetic macular edema
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SD-OCT Angiography (Experimental): Study participants will undergo imaging of both eyes with the AngioVue unit (approximately 60 seconds/eye), per standard operating protocol. Imaging is noncontact, and pharmacologic dilation will not be used for the purposes of this study. In most instances, study participants will undergo only a single imaging session on a single day. However, potential participants will be asked to consent for additional imaging sessions (up to 12) that may occur over the course of subsequent future visits to the clinic. Additionally, study participants will be asked to consent to prospective collection of clinical and demographic data, to correlate findings of OCT-A imaging to subsequent clinical course.
  Interventions: Device: AngioVue SD-OCT

INTERVENTIONS:
Device: AngioVue SD-OCT — OCT-A allows noninvasive, high-resolution imaging of the microvasculature of the retina and choroid, without intravenous dye administration. SD-OCT units use the light source used in commercially available and FDA-cleared OCT units on a modified platform. Optovue, Inc. has developed a customized SD-OCT system that implements a novel algorithm, the amplitude-based method of split-spectrum amplitude-decorrelation angiography (SSADA) for OCT-A. This detects motion in the blood vessel lumen by measuring the variation in reflected OCT signal amplitude between consecutive cross-sectional scans. Optovue has integrated the novel SSADA algorithm into their commercially approved RTVue SD-OCT unit for their OCT-A unit, the AngioVue. This unit is being conducted under an abbreviated IDE.

SUMMARY:
The objective of this study is to image retinal vascular alterations in patients with retinal disease using the AngioVue OCT-A system and understand the information these images provide. The investigators will image study participants who have retinal diseases with the AngioVue unit (Optovue) and will collect relevant clinical data to understand the nature of the information contained in images obtained on AngioVue. This study being conducted under an abbreviated IDE. The investigators will analyze data using descriptive statistics. Risks related to light exposure will be managed by ensuring that the exposure to the AngioVue light source is well below maximum permissible limits for safe exposure.

DETAILED DESCRIPTION:
OCT is an optical ranging and imaging technique first described in 1991 that has since been used successfully to provide high-resolution, micrometer-scale depth imaging in clinical ophthalmology (and other fields). It can be thought of as the optical analogue of ultrasound imaging. For the ocular posterior segment, OCT provides rapid acquisition of high-resolution, cross-sectional images of the retina that approximate tissue histology. In vivo imaging of the retina with OCT has thus dramatically improved clinicians' diagnostic capabilities, allowing earlier and more accurate diagnosis of disease and more precise assessment of response to therapies over time.

While OCT provides important information on retinal anatomy, it is currently limited in its ability to provide information on retinal vasculature and blood flow. Angiography is the current gold-standard imaging modality for retinal vascular imaging. Angiography involves intravenous injection of a fluorescent dye (typically either fluorescein or indocyanine green for the retinal or choroidal vessels, respectively) that circulates through the body. A light source emitting light at the specific excitation wavelength of the dye is placed in front of the patient's eye, and a camera equipped with a filter corresponding to the emission wavelength of the dye is then used to image vessel morphology and retinal perfusion, either through still images or through a short movie. Angiography provides physiologic information about the retina that complements the anatomical information provided by OCT. While generally well tolerated by most patients, angiography does have drawbacks: it often requires the use of a separate imaging system, it requires several minutes for image acquisition, and it involves intravenous injection of a dye. Patients occasionally experience side effects of intravenous dye administration, including nausea, discomfort, and rarely, anaphylaxis.

Several retinal imaging companies are developing the next generation of OCT technology: OCT angiography (OCT-A). OCT-A allows noninvasive, high-resolution imaging of the microvasculature of the retina and choroid (the vascular plexus subjacent to the retina), without the need for intravenous dye administration. OCT-A platforms currently under development include both spectral domain (SD) and swept-source (SS) based technologies. Whereas SS-based OCT-A utilizes a longer wavelength (~1060 nm) light source, SD-based units use the same light source used in commercially available and FDA-cleared OCT units on a modified platform. Optovue, Inc. (Fremont, CA) has developed one such unit, a customized, high-resolution SD-OCT system that implements a novel algorithm, the amplitude-based method of split-spectrum amplitude-decorrelation angiography (SSADA) for OCT-A. This SSADA algorithm allows for detection of motion in the blood vessel lumen by measuring the variation in reflected OCT signal amplitude between consecutive cross-sectional scans. Optovue has integrated the novel SSADA algorithm into their commercially approved RTVue SD-OCT unit for their OCT-A unit, the AngioVue. The AngioVue can generate high-quality angiograms of both the retina and choroid. Additionally, this refined method has produced images of the smallest retinal vessels (capillaries) in normal healthy control participants. In this proposed prospective interactive clinical study, we will use the AngioVue unit to image patients and characterize vascular abnormalities that are present in the setting of retinal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide consent
* History of clinically diagnosed retinal diseases, including but not limited to age-related macular degeneration, diabetic retinopathy, retinal vein occlusion, macular telangiectasias, and diabetic macular edema
* At least 18 years of age

Exclusion Criteria:

* Unable or unwilling to give consent
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-07; Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priyatham Mettu, MD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SD-OCT Angiography: Study participants will undergo imaging of both eyes with the AngioVue unit (approx. 60 seconds/eye), per standard operating protocol. Imaging is noncontact, and pharmacologic dilation will not be used for the purposes of this study. In most instances, study participants will undergo only a single imaging session on a single day. However, potential participants will be asked to consent for additional imaging sessions (up to 12) that may occur over the course of subsequent future visits to the clinic. Additionally, study participants will be asked to consent to prospective collection of clinical and demographic data, to correlate findings of OCT-A imaging to subsequent clinical course.
  AngioVue SD-OCT: OCT-A allows noninvasive, high-resolution imaging of the microvasculature of the retina and choroid, without intravenous dye administration. SD-OCT units use the light source used in commercially available and FDA-cleared OCT units on a modified platform. Optovue, Inc. has developed a customized SD-OCT system that implements a novel algorithm, the amplitude-based method of split-spectrum amplitude-decorrelation angiography (SSADA) for OCT-A. This detects motion in the blood vessel lumen by measuring the variation in reflected OCT signal amplitude between consecutive cross-sectional scans. Optovue has integrated the novel SSADA algorithm into their commercially approved RTVue SD-OCT unit for their OCT-A unit, the AngioVue. This unit is being conducted under an abbreviated IDE.
Period: Overall Study
Arm/Group | SD-OCT Angiography
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SD-OCT Angiography
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Image Quality Sensitive Enough to Identify Specific New Vessel Morphology
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Groups:
- SD-OCT Angiography: Study participants will undergo imaging of both eyes with the AngioVue unit (approx 60 seconds/eye), per standard operating protocol. Imaging is noncontact, and pharmacologic dilation will not be used for the purposes of this study. In most instances, study participants will undergo only a single imaging session on a single day. However, potential participants will be asked to consent for additional imaging sessions (up to 12) that may occur over the course of subsequent future visits to the clinic. Additionally, study participants will be asked to consent to prospective collection of clinical and demographic data, to correlate findings of OCT-A imaging to subsequent clinical course.
  AngioVue SD-OCT: OCT-A allows noninvasive, high-resolution imaging of the microvasculature of the retina and choroid, without intravenous dye administration. SD-OCT units use the light source used in commercially available and FDA-cleared OCT units on a modified platform. Optovue, Inc. has developed a customized SD-OCT system that implements a novel algorithm, the amplitude-based method of split-spectrum amplitude-decorrelation angiography (SSADA) for OCT-A. This detects motion in the blood vessel lumen by measuring the variation in reflected OCT signal amplitude between consecutive cross-sectional scans. Optovue has integrated the novel SSADA algorithm into their commercially approved RTVue SD-OCT unit for their OCT-A unit, the AngioVue. This unit is being conducted under an abbreviated IDE.
Arm/Group | SD-OCT Angiography
Number analyzed (Participants) | 39
Participants | 39

ADVERSE EVENTS:
Time Frame: Day 0
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | SD-OCT Angiography
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT02510885/Prot_SAP_000.pdf